CLINICAL TRIAL: NCT01618734
Title: Eltrombopag and Romiplostim Used Alternatively in Patients With Immune Thrombopenia (ITP).
Brief Title: Eltrombopag and Romiplostim Used Alternatively in Patients With Immune Thrombopenia (ITP): Efficacy and Safety.
Status: Completed | Type: Observational
Sponsor: Henri Mondor University Hospital (Other)
Collaborators: Paris 12 Val de Marne University (Other)
Responsible Party: Principal Investigator, Khellaf Mehdi, Medical Doctor, Henri Mondor University Hospital
Other Study IDs: TPO-r switch; TPO-r Switch in ITP
Record Dates: First submitted 2012-06-11; First posted 2012-06-13 (Estimated); Last update posted 2012-06-13 (Estimated); Status verified 2012-06

CONDITIONS: Immune Thrombocytopenia; Thrombopoietin Receptor Agonist
Keywords: Immune Thrombocytopenia; Thrombopoietin receptor agonist
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Romiplostim and eltrombopag in ITP: ITP patients who received alternatively romiplostim or eltrombopag with at least two months of follow-up for each period.

SUMMARY:
TPO-r Switch is a retrospective study of the patients affected by Immune Thrombopenia (ITP) who received alternatively romiplostim and eltrombopag.

DETAILED DESCRIPTION:
Thrombopoietin mimetics agents are available since 5 years in France through clinical trials first and then after their license. Two drugs are used: romiplostim and eltrombopag. These molecules have the same receptor on the megacaryocyte and induce the same stimulation of this cell leading to the differentiation and the proliferation into platelets. But romiplostim and eltrombopag have 2 different characteristics: the way of administration (oral for eltrombopag and subcutaneous for romiplostim) and the binding site to the C-MPL receptor on megacaryocyte. The aim of this study is to describe ITP patients who received these two drugs alternatively in order to know if there is a benefit for switching these molecules in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Subject has a diagnosis of ITP according to the American Society of Hematology guidelines (Rodeghiero et al, 2009).
* Subject is equal to or greater than 18 years of age.
* Before any study-specific procedure, the appropriate written informed consent must be obtained.
* Subject receiving romiplostim and eltrombopag alternatively
* Available follow-up of 2 months at least for each period

Exclusion Criteria:

- Secondary ITP e.g: thrombopenia related to hepatitis C, HIV, Chronic Lymphocytic Leukemia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with primary Immune Thrombopenia receiving romiplostim and eltrombopag alternatively.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2012-01; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Rate of efficacy after switching from one TPO mimetics to a second one. | 2 months minimun
  The primary outcome of this study is to know if switching from one TPO mimetics to a second one in ITP patients lead to a better efficacy in a significative proportion of patients.

SECONDARY OUTCOMES:
Rate of patients with an adverse events who have a benefit after switching. | 6 months
  Some ITP patients under TPO-r mimetics have some adverse events, the secondary outcome of this study is to evaluate the benefit to switch from one TPO-r mimetics to a second one in these cases.

REFERENCES:
- [Derived] Khellaf M, Viallard JF, Hamidou M, Cheze S, Roudot-Thoraval F, Lefrere F, Fain O, Audia S, Abgrall JF, Michot JM, Dauriac C, Lefort S, Gyan E, Niault M, Durand JM, Languille L, Boutboul D, Bierling P, Michel M, Godeau B. A retrospective pilot evaluation of switching thrombopoietic receptor-agonists in immune thrombocytopenia. Haematologica. 2013 Jun;98(6):881-7. doi: 10.3324/haematol.2012.074633. Epub 2013 Feb 26. PMID 23445876